CLINICAL TRIAL: NCT03585387
Title: Fluoroscopy vs Cardiac Positioning System Comparison to Assist the Navigation and Positioning of a Balloon Catheter in a Peripheral Artery During an Angioplasty Procedure
Brief Title: Cardiac Positioning System in Peripheral Angioplasty Procedure.
Acronym: MDG-Periph
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 10252
Record Dates: First submitted 2018-06-19; First posted 2018-07-13 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Main: Each subject in this group will be its own control for the two navigation methods.
  Interventions: Procedure: Navigation

INTERVENTIONS:
Procedure: Navigation — Navigation of a balloon catheter using two navigation methods (1-Fluoroscopy only; 2- Fluoroscopy + CPS).

SUMMARY:
This clinical investigation is intended to evaluate the ability of a magnetic cardiac positioning system to decrease medical radiation exposure on a peripheral angioplasty procedure in patients with a peripheral artery stenosis.

DETAILED DESCRIPTION:
The present study aims at addressing the fluoroscopy exposure time concern among physicians by proposing a new methodology that capitalizes on the cardiac positioning system (CPS) to reach near-zero fluoroscopy time for interventional cardiologists.

Intracoronary navigation of balloon catheter toward an anatomical landmark will be done with two navigation method:

1. Fluoroscopy alone
2. Fluoroscopy + CPS combination.

The order of the navigation method (method 1 then method 2 or vice versa) will be determine arbitrarily determined for each subject.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Scheduled for clinically indicated or contemplated percutaneous transluminal angioplasty or stenting of an peripheral artery;
* Able to provide informed consent for study participation and willing and able to comply with the Clinical Investigational Plan described evaluation.

Exclusion Criteria:

* Pregnant women or women planning to be pregnant during the study.
* Patients currently participating in another clinical study
* Patients with a thrombophilia
* Patients with critical limb ischemia
* Patients with unstable clinical condition or conditions limiting life expectancy that, in the opinion of the Study Investigator, excludes the participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective single-center, acute data collection study in 12 patients suffering from a peripheral arterial disease with an indication for an angioplasty procedure.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Time of radiation | Changes from time the balloon leaves the sheath to final alignment with anatomical landmark every 15 minutes over 2 hours.
  Medical radiation exposure for each balloon positioning

SECONDARY OUTCOMES:
Time duration | From time the balloon leaves the sheath to final alignment with anatomical landmark every 15 minutes over a 2 hours time frame.
  Procedure time for each balloon catheter positioning.
Dose area product (DAP) | DAP change from when balloon leaves the sheath to final alignment with anatomical landmark assessed every 15 minutes over a 2 hours time frame.
  Total amount of radiation delivered to the patient
Success or no-success in balloon navigation | Determined every 15 minutes over a 2 hours time frame.
  Physician assessment of balloon navigation and center alignment with an anatomical landmark.
Volume of contrast required to get the balloon to the anatomical landmark. | Change of volume of contrast from when balloon leaves the sheath to final alignment with anatomical landmark assessed every 15 minutes over a 2 hours time frame.
  Volume used
Distance measurements | At end of procedure
  Distance between the center of balloon aligned with anatomical landmark and the two radiopaque balloon markers.
Number of adverse events. | At end of procedure
  Adverse event count

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No